CLINICAL TRIAL: NCT06527547
Title: Effect of Transcutaneous Auricular Electroacupuncture on Sleep Disturbances in Patients With Rheumatoid Arthritis: A Randomized Double-Blind Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Jiao (Other)
Collaborators: Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Shenzhen Futian Hospital of TCM (Other Government); Inner Mongolia Autonomous Region Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Juan Jiao, professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-139-KY-01; CI2021B007 (Other Grant/Funding Number: Traditional Chinese Medicine Technology Innovation Team for Rheumatology)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-08

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Rheumatoid Arthritis; Sleep Quality
MeSH Terms: conditions — Arthritis, Rheumatoid; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- taVNS Group (Experimental): This arm consists of 26 participants diagnosed with rheumatoid arthritis who will receive transcutaneous auricular vagus nerve stimulation (taVNS) using the Huatuo electronic acupuncture device (model SDZ-IIB). Participants will be trained by a qualified physician to correctly position the earpieces on the auricular points corresponding to the heart and kidney. Treatment will be conducted at home, with each participant undergoing stimulation twice daily for 30 minutes each session, over a period of 5 consecutive days each week. The total intervention duration will last for 4 weeks. The stimulation frequency will be set at 20 Hz, using a sparse-dense wave pattern, with the intensity adjusted to the maximum level tolerated by the patient without causing pain.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Sham Stimulation Group (Sham Comparator): This arm includes 26 participants with rheumatoid arthritis who will receive sham stimulation using the same Huatuo electronic acupuncture device (model SDZ-IIB). Participants will be instructed on how to properly use the device, which will involve special sham electrodes placed over different ear areas not corresponding to therapeutic points (on the ear helix, specifically over the clavicle and shoulder points). The sham treatment will follow the same schedule as the experimental group: stimulation twice daily for 30 minutes per session, for 5 consecutive days each week, over 4 weeks. The device will be set to the same frequency and intensity as the experimental group, simulating the feeling of stimulation without delivering effective therapeutic intervention.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Treatment using the Huatuo electronic acupuncture device (model SDZ-IIB) with electrodes placed on the auricular points related to the heart and kidney. Pulsed wave type is sparse-dense wave, with a frequency of 20Hz and intensity set to the highest level tolerable without pain. Patients will perform self-treatment at home for 30 minutes, twice daily, for 5 days a week over 4 weeks.
  Arms: taVNS Group
Device: Sham Stimulation — Treatment using the same Huatuo electronic acupuncture device with electrodes placed on different ear points (over the ear helix). The device settings (pulse type, frequency, intensity) are the same as the experimental group but do not correspond to traditional acupuncture points. Patients will also perform self-treatment at home as per the same schedule as the experimental group.
  Arms: Sham Stimulation Group

SUMMARY:
The purpose of this clinical trial is to determine whether transcutaneous auricular vagus nerve stimulation (taVNS) is suitable for improving sleep disorders in patients with rheumatoid arthritis (RA). It will also evaluate the safety of taVNS. The main questions it aims to answer are:

Can taVNS improve the sleep quality of RA patients? What medical issues might RA patients experience while receiving taVNS treatment? Researchers will compare taVNS with a placebo (a similar substance that does not contain the actual treatment) to see if taVNS is effective in improving sleep disorders in RA patients.

Participants will:

Receive taVNS or sham stimulation daily for 4 weeks Keep a daily sleep diary and visit the hospital once a week for check-ups and tests Record their sleep quality and related symptoms This study aims to provide a new, safe, and effective non-drug therapy for sleep disorders related to RA.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the 2010 ACR/EULAR criteria for rheumatoid arthritis.
2. Poor sleep quality (PSQI score > 7).
3. Disease activity is moderate to low or in remission (DAS28 score ≤ 5.1).
4. No risk of sleep apnea (STOP-Bang questionnaire < 3).
5. Aged between 18 and 70.
6. The type and dosage of rheumatoid arthritis medication must be stable for at least 4 weeks.
7. Signed informed consent.

Exclusion Criteria:

1. People with acute infectious diseases, whether generalized or localized;
2. Those with severe internal organ diseases (such as coronary heart disease, arrhythmia, malignant tumors, renal failure, etc.);
3. Those working night shifts during the intervention period;
4. Those with other rheumatic diseases such as systemic lupus erythematosus, fibromyalgia, and Sjogren's syndrome;
5. Those undergoing treatment with steroids, sleeping pills, antidepressants, or antipsychotics;
6. Pregnant and breastfeeding women;
7. Those who cannot tolerate transcutaneous auricular electrostimulation.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index(PSQI) | Baseline, week1, week2, week3, week4
  Scores on the Pittsburgh Sleep Quality Index (PSQI) range from 0 to 21, with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
Consensus Sleep Diary-Core(CSD) | Baseline, week1, week2, week3, week4
  The Consensus Sleep Diary is primarily used to record and analyze sleep patterns and quality to help identify insomnia issues. While the Consensus Sleep Diary itself does not directly provide a scoring system, the recorded data can be used to calculate key sleep parameters. These parameters can be used to assess the severity of insomnia and the effectiveness of treatments.
Medical outcomes study sleep scale(MOS-SS) | Baseline,week4
  The MOS-SS Sleep Scale consists of 12 items and requires respondents to recall their sleep conditions over the past 4 weeks. Based on the scores for each item, the key indicators' scores are calculated.
Epworth sleepiness scale(ESS) | Baseline,week4
  The ESS consists of 8 questions, each describing a common daily activity. For each activity, respondents rate their tendency to doze off or fall asleep. The total score ranges from 0 to 24.
the Multidimensional Fatigue Inventory-20 (MFI-20) | Baseline,week4
  The Multidimensional Fatigue Inventory-20 (MFI-20) measures fatigue severity. The MFI-20 total score ranges from 0 to 80, with higher scores indicate more severe fatigue.
Tender joint count(TJC) | Baseline, week2, week4
  Tender Joint Count is a key clinical indicator in evaluating rheumatoid arthritis (RA). It measures the number of joints where patients feel pain upon touch or movement, helping to assess the disease's activity and severity. It involves 28 joints throughout the body.
Swollen joint count(SJC) | Baseline, week2, week4
  Swollen Joint Count (SJC) is another key clinical indicator for evaluating rheumatoid arthritis (RA). It measures the number of joints that are swollen due to inflammation, involving a total of 28 joints throughout the body.
Visual analogue scale(VAS) for pain | Baseline, week1, week2, week3, week4
  Pain VAS, range, 0 to 10 cm, where higher scores indicated the perceived pain to be more severe.
Disease Activity Score - 28 joints（DAS-28 ESR/CRP） | Baseline,week4
  DAS28 helps monitor RA progression, guide treatment, and is used in research. It provides a reliable measure for managing RA effectively.
Health Assessment Questionnaire（HAQ） | Baseline,week4
  The Health Assessment Questionnaire (HAQ) has a total of 20 items, each scored to reflect the patient's functional ability in daily life. The scores for each item are averaged, resulting in a total score ranging from 0 to 3.
Hospital Anxiety and Depression Scale（HADS） | Baseline,week4
  The Hospital Anxiety and Depression Scale (HADS) is a commonly used tool for screening and assessing anxiety and depression in general medical patients. The scale consists of 14 items. Each item is scored from 0 to 3 based on the severity of the symptoms, with a total score of 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No